CLINICAL TRIAL: NCT00506428
Title: Sleep, Aging, and Circadian Rhythm Disorders
Brief Title: Effects of Chronic Sleep Restriction in Young and Older People
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Institute on Aging (NIA) (NIH)
Responsible Party: Charles A Czeisler, PhD, MD, Brigham & Women's Hospital
Allocation: Non-Randomized | Model: Crossover | Masking: None
Other Study IDs: AG0077; 2P01AG009975-11 (NIH)
Record Dates: First submitted 2007-04-27; First posted 2007-07-25 (Estimated); Last update posted 2009-04-29 (Estimated); Status verified 2009-04

CONDITIONS: Aging; Sleep Deprivation; Metabolic Syndrome
Keywords: aging; sleep; sleep deprivation; performance; memory; metabolism
MeSH Terms: conditions — Sleep Deprivation; Metabolic Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: chronic sleep restriction — 5.6 hours of sleep per 24 hours for 3 weeks

SUMMARY:
The purpose of this study is to examine the consequences of chronic sleep restriction on nighttime sleep, daytime alertness, performance and memory functions, and metabolic and cardiovascular function, and to determine if the consequences of chronic sleep restriction differ between healthy young and older adults.

DETAILED DESCRIPTION:
It has long been recognized that sleep patterns change with age. A common feature of aging is the advance of the timing of sleep to earlier hours, often earlier than desired. Polysomnographically-recorded sleep in older people shows an increased number of awakenings, a reduction of stages 3 and 4 (SWS) sleep, and a flattening of REM sleep distribution throughout the night. These age-related changes are found in even healthy individuals who are not taking medications and who are free from sleep disorders. In addition to these sleep disturbances, many older individuals curtail their sleep voluntarily, reporting similar rates of sleep restriction (sleeping less than 7 or less than 6 hours per night) as young adults. Whether voluntary or not, insufficient sleep has medical, safety and metabolic consequences. In fact, converging evidence in young adults suggests that sleep restriction per se may impair metabolism, and that reduced sleep duration is associated with weight gain, obesity, diabetes, cardiovascular disease, and mortality.

The study begins with 21 days of outpatient study in which the participants will be required to sleep for 10 hours each night in order to ensure they are well-rested. This will be followed by a 39-day inpatient study. The study will begin with 3 "sleep satiation" days during which all participants will be scheduled to sleep for 12 hours per night and have a 4 hour nap each afternoon. This is followed by 3 baseline days in which the participants will follow the same sleep-wake schedule they were following at home. Following this, the participant will undergo 3 weeks of chronic sleep restriction while living on a non-24-hour schedule. The participant will live on a schedule that is equivalent to 5.6 hours of sleep per 24 hours. Following these 3 weeks, the participant will be scheduled to again sleep for 10 hours per night for 10 nights.

ELIGIBILITY:
Inclusion Criteria:

* Healthy

Exclusion Criteria:

* Chronic or acute medical condition
* Medication use
* Depression
* History of psychiatric illness
* Sleep disorder

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2006-12; Primary Completion 2011-06 (Estimated); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
Changes in sleep and waking EEG measures | During 3-week chronic sleep restriction segment of inpatient study
frequent measures of performance, attention, alertness, and memory | During 3-week chronic sleep restriction segment of inpatient study
measures of cardiovascular and metabolic function | During 3-week chronic sleep restriction segment of inpatient study

CONTACTS AND LOCATIONS:
Overall Officials: Charles A Czeisler, PhD, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham & Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Czeisler CA, Duffy JF, Shanahan TL, Brown EN, Mitchell JF, Rimmer DW, Ronda JM, Silva EJ, Allan JS, Emens JS, Dijk DJ, Kronauer RE. Stability, precision, and near-24-hour period of the human circadian pacemaker. Science. 1999 Jun 25;284(5423):2177-81. doi: 10.1126/science.284.5423.2177. PMID 10381883
- [Background] Dijk DJ, Duffy JF, Riel E, Shanahan TL, Czeisler CA. Ageing and the circadian and homeostatic regulation of human sleep during forced desynchrony of rest, melatonin and temperature rhythms. J Physiol. 1999 Apr 15;516 ( Pt 2)(Pt 2):611-27. doi: 10.1111/j.1469-7793.1999.0611v.x. PMID 10087357
- [Background] Dijk DJ, Shanahan TL, Duffy JF, Ronda JM, Czeisler CA. Variation of electroencephalographic activity during non-rapid eye movement and rapid eye movement sleep with phase of circadian melatonin rhythm in humans. J Physiol. 1997 Dec 15;505 ( Pt 3)(Pt 3):851-8. doi: 10.1111/j.1469-7793.1997.851ba.x. PMID 9457658
- [Background] Boivin DB, Czeisler CA, Dijk DJ, Duffy JF, Folkard S, Minors DS, Totterdell P, Waterhouse JM. Complex interaction of the sleep-wake cycle and circadian phase modulates mood in healthy subjects. Arch Gen Psychiatry. 1997 Feb;54(2):145-52. doi: 10.1001/archpsyc.1997.01830140055010. PMID 9040282
- [Background] Dijk DJ, Duffy JF, Czeisler CA. Circadian and sleep/wake dependent aspects of subjective alertness and cognitive performance. J Sleep Res. 1992 Jun;1(2):112-7. doi: 10.1111/j.1365-2869.1992.tb00021.x. PMID 10607036
- [Background] Duffy JF. Increased sleep disruption, reduced sleepiness in older subjects? Sleep. 2005 Nov;28(11):1358-9. No abstract available. PMID 16335324
- [Background] Klerman EB, Davis JB, Duffy JF, Dijk DJ, Kronauer RE. Older people awaken more frequently but fall back asleep at the same rate as younger people. Sleep. 2004 Jun 15;27(4):793-8. doi: 10.1093/sleep/27.4.793. PMID 15283016
- [Background] Duffy JF, Czeisler CA. Age-related change in the relationship between circadian period, circadian phase, and diurnal preference in humans. Neurosci Lett. 2002 Feb 1;318(3):117-20. doi: 10.1016/s0304-3940(01)02427-2. PMID 11803113
- [Background] Dijk DJ, Duffy JF, Czeisler CA. Age-related increase in awakenings: impaired consolidation of nonREM sleep at all circadian phases. Sleep. 2001 Aug 1;24(5):565-77. doi: 10.1093/sleep/24.5.565. PMID 11480654
- [Background] Dijk DJ, Duffy JF, Czeisler CA. Contribution of circadian physiology and sleep homeostasis to age-related changes in human sleep. Chronobiol Int. 2000 May;17(3):285-311. doi: 10.1081/cbi-100101049. PMID 10841208
- [Background] Pavlova MK, Duffy JF, Shea SA. Polysomnographic respiratory abnormalities in asymptomatic individuals. Sleep. 2008 Feb;31(2):241-8. doi: 10.1093/sleep/31.2.241. PMID 18274272
- [Background] Silva EJ, Duffy JF. Sleep inertia varies with circadian phase and sleep stage in older adults. Behav Neurosci. 2008 Aug;122(4):928-35. doi: 10.1037/0735-7044.122.4.928. PMID 18729646
- [Background] Munch MY, Cain SW, Duffy JF. Biological Rhythms Workshop IC: sleep and rhythms. Cold Spring Harb Symp Quant Biol. 2007;72:35-46. doi: 10.1101/sqb.2007.72.065. PMID 18419261
- [Derived] Swanson CM, Shea SA, Kohrt WM, Wright KP, Cain SW, Munch M, Vujovic N, Czeisler CA, Orwoll ES, Buxton OM. Sleep Restriction With Circadian Disruption Negatively Alter Bone Turnover Markers in Women. J Clin Endocrinol Metab. 2020 Jul 1;105(7):2456-63. doi: 10.1210/clinem/dgaa232. PMID 32364602
- [Derived] Swanson CM, Shea SA, Wolfe P, Cain SW, Munch M, Vujovic N, Czeisler CA, Buxton OM, Orwoll ES. Bone Turnover Markers After Sleep Restriction and Circadian Disruption: A Mechanism for Sleep-Related Bone Loss in Humans. J Clin Endocrinol Metab. 2017 Oct 1;102(10):3722-3730. doi: 10.1210/jc.2017-01147. PMID 28973223